CLINICAL TRIAL: NCT05275049
Title: Translingual Stimulation Combined With Physiotherapy to Improve Walking and Balance in Multiple Sclerosis: an RCT
Brief Title: Neuromodulation in MS Using Translingual Stimulation
Acronym: NeuroMSTraLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Saskatchewan (Other)
Collaborators: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Sarah Donkers, Principal Investigator, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio 2578
Record Dates: First submitted 2021-11-28; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: physiotherapy; walking and balance; neurorehabilitation; non-invasive cranial nerve neuromodulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PT+ Device (Experimental): PT plus translingual stimulation device PoNS device will be used to deliver trans-lingual electrical stimulation. The stimulation will be delivered while the participants engages in evidence-based physiotherapy for walking and balance.
  Interventions: Combination Product: PT plus translingual stimulation device
- PT + Control Device (Active Comparator): PT plus translingual stimulation control device Control device will be used. Participants will wear device while engaging in evidence-based physiotherapy for walking and balance.
  Interventions: Combination Product: PT plus translingual stimulation control device

INTERVENTIONS:
Combination Product: PT plus translingual stimulation device — PoNS device will be used to deliver trans-lingual electrical stimulation. The stimulation will be delivered while the participants engages in evidence-based physiotherapy for walking and balance.
  Arms: PT+ Device
Combination Product: PT plus translingual stimulation control device — Control device will be used. Participants will wear device while engaging in evidence-based physiotherapy for walking and balance.
  Arms: PT + Control Device

SUMMARY:
The overarching aim of this study is to examine if there is additional benefit to adding trans-lingual electrical stimulation to physiotherapy aimed at improving walking and balance in people with multiple sclerosis (MS).

DETAILED DESCRIPTION:
This is a two arm, participant-blinded, interventionist blinded, and research assessor-blinded RCT Participants with walking problems due to MS (Patient Determined Disease Steps PDDS 3-6) will be randomized 1:1 after baseline assessment stratified into 2 arms (lower walking disabilities PDDS 3+4, and higher walking disabilities PDDS 5+6) Following a 14 week balance and walking training intervention, participants will be instructed to continue to exercise independently according to the evidence-based Physical Activity Guidelines in MS for a subsequent 12 weeks. They will be reassessed at the end of that time (FOLLOW-UP).

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of multiple sclerosis
* gait deficit due to MS but still able to walk (EDSS less than 6.5, PDDS 3-6)
* older than 18 and less than 70 years of age
* agree to the study time commitment.

Exclusion Criteria:

* currently attending physical rehabilitation for walking and/or balance training,
* currently already functional community ambulators (gait speed>120cm/s)
* contra-indications to the use of translingual electrical stimulation (active or suspected malignant tumor; recent bleeding or open wounds in mouth; women who are pregnant, or sensitivity to nickel, gold or copper)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-07-05 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Timed 25 foot walk test (T25FWT) | 27 weeks
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. Time to complete the T25FWT, and walking seed will be calculated. A lower time and faster walking speed indicates better walking performance
Dynamic Gait Index (DGI) | 27 weeks
  This scale has 8 conditions that an individual walks in (e.g. normal, head turns, change in speed, pivot, stairs). Performance for each condition is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best score on the DGI is 24, and a higher score means less walking impairment.

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale (MSIS-29) | 27 weeks
  This is a 29 item self-reported questionnaire - 20 items deal with physical state and 9 with psychological. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where a larger number (e.g. closer to 100) indicates greater impact of disease on daily function.
Fatigue Scale for Motor and Cognitive Functions | 27 weeks
  This is a 20-item self-reported questionnaire, a Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made as 10 questions relate to motor fatigue and 10 to cognitive fatigue. A higher score means the individuals is more affected by fatigue.
Short From 36 Health Survey Questionnaire (SF-36) | 27 weeks
  This is a self-reported questionnaire used to rate health related quality of life. Eight health concepts are covered in 36 questions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The 36 items are rated using a number of different scales and an intricate formula is used to calculate a final score. A high score defines a more favorable health state
Multiple sclerosis walking scale - 12 item (MSWS-12) | 27 weeks
  This is a 12 item self-reported questionnaire where participants rate each item from 1-5, giving a total out of 60, and then transforming this to a scale with a range from 0 to 100%.
  Higher scores indicate a greater impact on walking than lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Donkers, Principal Investigator — University of Saskatchewan; Michelle Ploughman, Principal Investigator — Memorial University of Newfoundland
Locations (2):
- Canada (2):
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - University of Saskatchewan, Saskatoon, Saskatchewan